CLINICAL TRIAL: NCT04317833
Title: A Single Dose Escalation Study to Investigate the Tolerability, Safety, Pharmacokinetics and Pharmacodynamics of SSS17 in Chinese Healthy Subject
Brief Title: A Study of SSS17 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYSS-SSS17-UND-I-01
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Anemia in Chronic Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation SSS17 (Experimental): Escalating doses of SSS17; single dose administration; different dosage forms (redosing of the SSS17 in one cohort with food on Day15)
  Interventions: Drug: SSS17
- Escalation matching Placebo (Placebo Comparator): Escalating doses of matching placebo; single dose administration; different dosage forms (redosing of matching placebo in one cohort with food on Day15)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SSS17 — SSS17 is a novel small molecule compound which stimulates erythropoiesis through inhibition of hypoxia-inducible factor- prolyl hydroxylases( HIF-PH). It is being developed for the treatment of anemia in patients with chronic kidney disease.
  Arms: Dose Escalation SSS17
Drug: Placebo — matched placebo
  Arms: Escalation matching Placebo

SUMMARY:
This is a first-in-human, Phase 1, single-center, randomized, single-blind, placebo-controlled, single dose-escalation study to evaluate the safety, tolerability, PK, PD of SSS17 following oral administration in healthy subjects. Approximately 65 subjects (53 receiving active drug and 12 receiving placebo) will participate in this study.

DETAILED DESCRIPTION:
The study will enroll healthy volunteers from a single academic medical center in China. All participants will be informed about the study and potential risks and required to provide written informed consent prior to undergoing study-related procedures.

The improved Fibonacci dose escalation design will be implemented. The protocol specifies 10 mg, oral, one time for the first cohort without placebo control. Successive cohorts will be given doses up to 540 mg with placebo parallel control. Only no observation meets the criteria under stop rules, dose will escalate to the next higher level.

The study will be divided into 2 stages: 1st period (fast) and 2nd period(fed).

First period (fast): Subjects will be allocated 1:4 to receive placebo or SSS17, which will be administered by oral route. At each dose, tolerability, safety, PK and PD characteristics will be investigated.

Second period (fed): in order to investigate the effects of food on PK and PD of SSS17. Subjects in one cohort will be administered again after meal on Day15. The accurate dose will be adjusted according to the findings in 1st period (fast)

ELIGIBILITY:
Inclusion Criteria:

* Body weight≥50 for male or ≥45 for female, and BMI between 19.0-26.0 kg/m2
* Good general health as determined by the investigator based on medical history, physical examination, vital signs, 12-lead ECG, clinical laboratory tests and B-type ultrasound test.
* Participants of reproductive potential must agree to utilize reliable methods of contraception from screening to 6 months after the last administration of the study intervention. No plan for sperm (or egg) donation or pregnancy.
* Understand and sign the informed consent.
* Ability to understand and follow study-related instruction

Exclusion Criteria:

* A known allergy to any component of the SSS17 formulation, or allergy history of two kinds of drugs or food
* Medical history or conditions of digestive system.
* Female volunteers who are pregnant, menstrual, lactating or menopause with hormone therapy.
* Eyes diseases, including diabetic retinopathy, age-related macular degeneration.
* Vascular anomalies.
* Drug, alcohol or nicotine addiction.
* Blood donation or bleeding (more than 200 ml). Experience of treatment with EPO or blood transfusion.
* Any findings from the medical examination (including medical history, physical examination, vital signs, laboratory tests and ECG) deviating from normal and deemed by the investigator to be of clinical relevance
* Abnormal results in test of TIBC, serum iron or ferritin
* Acute diseases before administration.
* Other situations that the researcher believes may affect validity judgment or are not suitable for participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
AEs | up to Day14 or 29
  assessment AEs by frequency, severity

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of SSS17 | [ up to 48 hours post-dose]
  Plasma samples will be collected and Cmax will be assessed.
Area under the concentration-time curve (AUC) of plasma concentration of SSS17 | [ up to 48 hours post-dose]
  Plasma samples will be collected and the AUC from zero to infinity will be assessed.
Time-to-Cmax (Tmax) of SSS 17 | [ up to 48 hours post-dose]
  Plasma samples will be collected and the Tmax will be assessed from the concentration-time curve.
Elimination terminal half-life (t1/2) of SSS17 | [up to 48 hours post-dose]
  Plasma samples will be collected and the t1/2 will be assessed.
Total amount of SSS17 excreted in urine over 24 hours (Ae0-24) | only for one cohort (up to 72 hours post-dose)
  Urine sample will be collected at pre-specified intervals and Ae0-24 will be assessed.
Fraction of SSS17 excretion during each collection interval (Fe0-24) | only for one cohort (up to 72 hours post-dose)
  Urine sample will be collected at pre-specified intervals and Fe0-24 will be assessed.
Total amount of SSS17 excreted in urine over 72 hours (Ae0-72) | only for one cohort (up to 72 hours post-dose)
  Urine sample will be collected at pre-specified intervals and Ae0-72 will be assessed.
Fraction of SSS17 excretion during each collection interval (Fe0-72) | only for one cohort (up to 72 hours post-dose)
  Urine sample will be collected at pre-specified intervals and Fe0-72 will be assessed.
Renal clearance (CLR) of SSS17 | only for one cohort (up to 72 hours post-dose)
  Urine sample will be collected at pre-specified intervals and CLR will be assessed.
EPO concentrations | up to 168 hours post-dose.
  Change of EPO concentrations from baseline following SSS17
VEGF concentrations | up to 168 hours post-dose.
  Change of VEGF concentrations from baseline following SSS17
Change of RTC from baseline | up to 168 hours post-dose.
  Change of RTC from baseline following SSS17
Change of RBC from baseline | up to 168 hours post-dose.
  Change of RBC from baseline following SSS17
Change of Hgb from baseline | up to 168 hours post-dose.
  Change of Hgb from baseline following SSS17
Change of hepcidin from baseline | up to 168 hours post-dose.
  Change of serum hepcidin concentrations from baseline following SSS17

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided